CLINICAL TRIAL: NCT02453100
Title: Managing Urinary Incontinence in Elderly Village Women in Rural Bangladesh: a Cluster Randomized Trial of a Community Exercise-based Intervention
Brief Title: Managing Urinary Incontinence in Elderly Village Women in Rural Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Gonoshasthaya Kendra Bangladesh (Unknown)
Responsible Party: Principal Investigator, Nicola Cherry, Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RES0022238
Record Dates: First submitted 2015-05-19; First posted 2015-05-25 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Range of Motion, Articular; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): Women will be included in group mobility and pelvic floor exercise classes for one and a half hours twice weekly for 12 weeks and encouraged to carry out independent exercises each day when there is no group session.
  A research paramedics will meet with the woman each month for six months from the initial training session to encourage her continued participation and adherence to the individual exercise program. At this meeting the research paramedic will also provide and reinforce simple education about how to manage urinary incontinence.
  Interventions: Behavioral: Mobility and pelvic floor exercise; Behavioral: Education
- Education (Placebo Comparator): On recruitment and each month for six months a research paramedic will meet with each woman to provide and reinforce simple education about how to manage urinary incontinence.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Mobility and pelvic floor exercise — Mobility and pelvic floor exercises
  Arms: Exercise
Behavioral: Education — Education on simple ways to manage incontinence

SUMMARY:
An intervention consisting of group and home based exercise will be used over 6 months to assess whether this is helpful in managing urinary incontinence in elderly village women in Bangladesh. This intervention, supplemented by education about managing incontinence, will be used in half the villages in the trial. In the other half women will receive only the education component.

DETAILED DESCRIPTION:
This is a cluster randomized trial in which all women aged 60-75 years reporting symptoms of urinary incontinence are randomly assigned, by village of residence, to either exercise plus education of to education alone.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 60-75 years reporting incontinence on a screening questionnaire (yes to questions 2,3or 4 on the 6 item Urinary Distress Index)

Exclusion Criteria:

* They report a uterine prolapse which is (or becomes) known to be of 3rd degree or higher.
* They are assessed by the village paramedic to be incapable of standing from sitting without help from someone else.
* They are assessed by the village paramedic to be unable to walk without help at a normal pace for someone of her age.
* They are assessed by the village paramedic as not having the intellectual capacity to understand questions and follow instructions.

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 579 (Actual)
Dates: Start 2015-06; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Frequency of involuntary leakage of urine | Baseline and 24 weeks
  The frequency of involuntary leakage over 3 days will be measured at each time point

SECONDARY OUTCOMES:
Frequency of micturition | Baseline and 24 weeks
  The frequency of micturition over 3 days will be measured at each time point
Severity of urinary symptoms | Baseline, 12 weeks and 24 weeks
  Urinary symptoms measured by the 2 item Sandvick index of severity
Depression as measured on a Bangla version of the 10 item Center for Epidemiological Studies Depression Scale (CES-D 10) | Baseline, 12 weeks and 24 weeks
  Depression as measured on a Bangla version of the CES-D 10
Quality of life as measured by a Bangla version of the Euroqol 5 dimension scale (EQ-5D) | Baseline and 24 weeks
  Quality of life as measured by a Bangla version of the EQ-5D
Distress caused by urinary symptoms | Baseline and 24 weeks
  Distress measured by the 6 item Urinary Distress Index

CONTACTS AND LOCATIONS:
Overall Officials: Nicola M Cherry, MD PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Wagg A, Chowdhury Z, Galarneau JM, Haque R, Kabir F, MacDonald D, Naher K, Yasui Y, Cherry N. Exercise intervention in the management of urinary incontinence in older women in villages in Bangladesh: a cluster randomised trial. Lancet Glob Health. 2019 Jul;7(7):e923-e931. doi: 10.1016/S2214-109X(19)30205-0. PMID 31200891